CLINICAL TRIAL: NCT02747459
Title: Sensory Supported Swimming-Swimming and Water Safety for Children With Autism Spectrum Disorder
Brief Title: Sensory Supported Swimming for Children With ASD
Acronym: SSS
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Lisa Mische Lawson, PhD, Associate Professor, University of Kansas Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 13124
Record Dates: First submitted 2016-04-19; First posted 2016-04-21 (Estimated); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Autism Spectrum Disorders
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SSS Intervention (Experimental): Sensory Supported Swimming-eight, 30 minute lessons
  Interventions: Behavioral: Sensory Supported Swimming

INTERVENTIONS:
Behavioral: Sensory Supported Swimming — A swimming and water safety program for children with autism spectrum disorders. Individualized instruction utilizing evidence-based teaching methods and sensory modifications.
  Other Names: Sensory Enhanced Aquatics

SUMMARY:
The purpose of Sensory Supported Swimming is to provide a sustainable, low cost recreational swim program for children with ASD. A secondary purpose is to train general recreation providers and swim instructors to meet the unique needs of children. Specific aims include both program development and research aims as described below.

Specific Aims:

1. Provide more opportunities for families of children with ASD to access a recreational swim program at low cost. (program development) 2. Increase the capacity of swim instructors and general recreation providers working with children with ASD. (Research) 3. Increase physical activity for children with ASD in a way that is a good match for their individual sensory needs. (Research) 4. Increase safety among children with ASD in and around the water so they and their families can swim safely. (Research) 5. Transition swimmers with ASD from a learn-to-swim program to an inclusive swim team. (Program Development) Hypotheses

1. The Sensory Supported Swim Program will increase physical activity of children with ASD.
2. The Sensory Supported Swim Program will increase safety of children with ASD in and around the water.
3. The Sensory Supported Swim Program will increase the capacity of general recreation providers and swim instructors to serve children with ASD.

DETAILED DESCRIPTION:
To decrease risk of drowning, increase opportunities to engage in a lifelong sport, and increase the capacity of general recreation providers, investigators developed a recreational swim program for children with ASD. The purpose of this program is to provide swimming and water safety instruction for children with ASD. A secondary purpose is to train general recreation providers and swim instructors to meet the unique needs of children. Research of this program includes investigating the effects of swimming on health outcomes (i.e., fitness, BMI) of children with ASD. SSS lessons are provided in eight week sessions six times per year. Lessons are individualized according to the child's sensory preferences (as measured by the Sensory Profile). Instructors use evidence-based teaching methods (i.e., visual supports, demonstration, peer and video modelling, sensory modifications) to teach swimming and water safety skills. Children may enroll for as many sessions as desired. Research includes retrospective review of program records.

ELIGIBILITY:
Inclusion Criteria:

* Autism diagnosis (any autism spectrum diagnosis)
* Order of response

Exclusion Criteria:

* Children with sensory impairments (i.e., blindness, deafness)
* Based on the discretion of the program directors, participants that display aggressive or harmful behaviors may be excluded for safety purposes

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 500 (Estimated)
Dates: Start 2012-03; Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Skill Acquisition Form | 8 weeks
  This outcome measure was created for the study to measure changes in swimming and water safety skills. The skill acquisition form is supplemented with weekly progress notes.

SECONDARY OUTCOMES:
Instructor Survey | 16 weeks
  Instructors are surveyed at least annually to determine if Sensory Supported Swimming is increasing their competence to serve children with autism spectrum disorders
Parent Survey | 16 weeks
  Parents of program participants are surveyed at least annually to determine if Sensory Supported Swimming is increasing children's physical activity and safety around water
Program Records | 8 weeks
  demographics forms, enrollment & attendance records

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Mische Lawson, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No
Data is only used my KUMC study team

REFERENCES:
- [Derived] Lawson LM, Foster L. Sensory Patterns, Obesity, and Physical Activity Participation of Children With Autism Spectrum Disorder. Am J Occup Ther. 2016 Sep-Oct;70(5):7005180070p1-8. doi: 10.5014/ajot.2016.021535. PMID 27548863